CLINICAL TRIAL: NCT07172139
Title: Effect of Transcranial Magnetic Stimulation vs Sham Stimulation Combined With Pinaverium Bromide vs Bifidobacteria in Diarrhea-Predominant Irritable Bowel Syndrome: A 2×2 Factorial Randomized Clinical Trial
Brief Title: Transcranial Magnetic Stimulation and Pharmacologic/Probiotic Interventions for Diarrhea-Predominant IBS
Acronym: rTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rui Li (Other)
Responsible Party: Sponsor-Investigator, Rui Li, The First Affiliated Hospital of Soochow University, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2025655
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: IBS (Irritable Bowel Syndrome)
Keywords: Diarrhea-predominant Irritable Bowel Syndrome; repetitive Transcranial Magnetic Stimulation; Pinaverium Bromide; Bifidobacterium; chronic visceral pain
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — pinaverium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent researcher will generate a randomized sequence using an online tool (https://www.sealedenvelope.com/simple-randomiser/v1/lists) with 1:1:1:1 allocation stratified by center. The attending physician will open sealed envelopes before treatment to assign participants to one of four groups: rTMS with pinaverium, rTMS with Bifidobacterium, sham with pinaverium, or sham with Bifidobacterium. Block randomization (block size=4) ensures balance across centers.
  For blinding, identical capsules conceal medications from patients and outcome assessors. Participants are blinded to real/sham rTMS due to identical auditory cues. rTMS operators are unblinded but excluded from outcome assessment. All other personnel remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active rTMS + Pinaverium Bromide Group (Experimental): Participants in this arm will receive active repetitive Transcranial Magnetic Stimulation (rTMS) sessions and oral Pinaverium Bromide tablets.
  Interventions: Combination Product: Active rTMS + Pinaverium Bromide
- Active rTMS + Bifidobacterium Group (Experimental): Participants in this group will receive active repetitive Transcranial Magnetic Stimulation (rTMS) sessions and oral Bifidobacterium supplements.
  Interventions: Combination Product: Active rTMS + Bifidobacterium
- Sham rTMS + Pinaverium Bromide Group (Sham Comparator): Pinaverium Bromide 50 mg film-coated tablets. Administered orally at a dosage of 50 mg (one tablet) three times daily, 30 minutes before meals, for a duration of 2 weeks.
  Interventions: Combination Product: Sham Comparator: Sham rTMS + Pinaverium Bromide
- Sham rTMS + Bifidobacterium Group (Placebo Comparator): Each capsule contains a minimum of 5 billion colony-forming units (CFU). Administered orally at a dosage of one capsule twice per day, with meals, for a duration of 2 weeks. The product will be stored refrigerated as per manufacturer's instructions.
  Interventions: Combination Product: Placebo Comparator: Sham rTMS + Bifidobacterium

INTERVENTIONS:
Combination Product: Active rTMS + Pinaverium Bromide — A figure-of-eight coil is used to apply active low-frequency (1 Hz) rTMS to the corresponding representation area of the prefrontal cortex (mPFC). The treatment is administered for 20 minutes daily for a total of 2 weeks.
  Arms: Active rTMS + Pinaverium Bromide Group
Combination Product: Active rTMS + Bifidobacterium — Bifidobacterium animalis subsp. lactis BB-12, provided in capsule form. Each capsule contains a minimum of 5 billion colony-forming units (CFU). Administered orally at a dosage of one capsule twice per day, with meals, for a duration of 2 weeks. The product will be stored refrigerated as per manufacturer's instructions.
  Arms: Active rTMS + Bifidobacterium Group
Combination Product: Sham Comparator: Sham rTMS + Pinaverium Bromide — Pinaverium Bromide 50 mg film-coated tablets. Administered orally at a dosage of 50 mg (one tablet) three times daily, 30 minutes before meals, for a duration of 2 weeks.
  Arms: Sham rTMS + Pinaverium Bromide Group
Combination Product: Placebo Comparator: Sham rTMS + Bifidobacterium — Description: Sham stimulation is delivered using a placebo coil that mimics the sound and sensation of active rTMS but does not deliver the full magnetic field. Parameters identical to active arm.
  Arms: Sham rTMS + Bifidobacterium Group

SUMMARY:
What is the study about? This study is for adults with diarrhea-predominant irritable bowel syndrome (IBS-D) who suffer from chronic visceral pain. We aim to investigate whether combining two different treatment approaches is more effective in alleviating IBS-D symptoms than either treatment alone. The first treatment is a non-invasive brain stimulation technique called repetitive Transcranial Magnetic Stimulation (rTMS), while the second treatment involves either an intestinal antispasmodic medication (Pinaverium Bromide) or a probiotic (Bifidobacterium).

What will participants do?

Participants will be randomly assigned by a computer to one of four groups:

1. Group 1: Receive real rTMS sessions + take Pinaverium Bromide pills.
2. Group 2: Receive real rTMS sessions + take Bifidobacterium pills.
3. Group 3: Receive fake (sham) rTMS sessions + take Pinaverium Bromide pills.
4. Group 4: Receive fake (sham) rTMS sessions + take Bifidobacterium pills.

Neither the participant nor the doctor giving the treatments will know which group the participant is in for the rTMS part (this is called "blinding"). The study will involve several weeks of treatment and follow-up visits to track symptoms.

What are the potential benefits and risks? Potential Benefits: Participants may experience a reduction in their abdominal pain, diarrhea, and other IBS symptoms. However, benefit cannot be guaranteed. The information from this study may help other IBS patients in the future.

Potential Risks: rTMS is generally safe but may cause mild headache, scalp discomfort, or lightheadedness. The medications may have side effects like any drug, which will be explained in detail before the study starts.

Why is this study important? This is the first study to test how brain stimulation and gut-focused treatments work together for IBS pain. The results could lead to new and more effective combination therapies for people who don't get enough relief from current treatments.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, sham-controlled, 2x2 factorial trial investigating the efficacy of combining repetitive Transcranial Magnetic Stimulation (rTMS) with gut-directed therapy for chronic visceral pain in diarrhea-predominant irritable bowel syndrome (IBS-D).

Scientific rationale: Current treatments for IBS-D often provide inadequate relief. rTMS, a non-invasive neuromodulation technique, may alleviate pain by restoring cortical excitability and neural plasticity. Its potential synergy with gut-targeted agents (antispasmodic or probiotic) remains unexplored.

Objectives: The primary objective is to determine the interaction effect between rTMS (real vs. sham) and drug (pinaverium bromide vs. bifidobacterium) on the composite response rate at Week 2. Secondary objectives include assessing changes in IBS-SSS, IBS-QoL, PHQ-9 scores, and anorectal manometry parameters.

Methodology: 140 eligible adults will be randomized equally into four groups: (1) real rTMS + pinaverium bromide, (2) real rTMS + bifidobacterium, (3) sham rTMS + pinaverium bromide, (4) sham rTMS + bifidobacterium. Real rTMS will be delivered at 1Hz, 80% MT over the mPFC for 20 minutes daily for 2 weeks. Sham rTMS uses a placebo coil. Pinaverium bromide (50mg tid) and bifidobacterium (500mg bid) will be administered with matched placebos to maintain blinding. Participants, outcome assessors, and statisticians will be blinded to intervention assignments.

Outcomes: The primary outcome is the proportion of participants achieving composite response (≥30% reduction in worst abdominal pain AND ≥50% reduction in days with BSFS 6/7 stools) at Week 2. Secondary outcomes include changes from baseline in IBS-SSS, IBS-QoL, PHQ-9, and manometry measures.

Statistics: A factorial ANOVA will be used to test the main and interaction effects. The primary analysis will follow the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

(I)Age range 18-75 years (either sex) (II)Fulfilling the Rome IV criteria for irritable bowel syndrome diagnosis (III)Bristol stool type 6-7 in >25% and type 1-2 in <25% of bowel movements (IV)Patients experienced Bristol stool type 6 or 7 on ≥4 days with mean abdominal pain score ≥3 during the initial 2-week period

Exclusion Criteria:

(I)Documented organic gastrointestinal pathology; endocrinologic or metabolic diseases with known gastrointestinal motility effects including diabetes mellitus and hyperthyroidism; previous surgical interventions involving abdominal cavity intestinal tract or anal region (II)current use of any medication with documented effects on gastrointestinal motility or secretory function; administration of concurrent therapies or pharmacologic agents capable of confounding treatment efficacy or safety evaluations (III)pregnancy lactation or postpartum status within 12 months (IV)noncompliance with randomized treatment allocation or demonstrated poor adherence tendencies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with composite response | At Week 2 (end of treatment)
  The primary outcome measure is the proportion of patients achieving a composite response at the end of treatment (Week 2), defined as: a reduction of ≥30% from baseline in the average daily worst abdominal pain score, and a reduction of ≥50% in the number of days with at least one stool consistency meeting BSFS type 6 or 7 criteria during Week 2. Abdominal pain intensity is assessed using an 11-point NRS scale (0-10) for the last 24 hours daily. Stool consistency is recorded daily by the patient selecting the most representative category according to the BSFS.

SECONDARY OUTCOMES:
Symptoms, Quality of Life | From baseline to week 2 of treatment
  The IBS Symptom Severity Scale (IBS-SSS) is utilized to assess the overall symptomatology of irritable bowel syndrome. This scale comprises five domains: severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and impact on quality of life. Each domain is scored on a scale from 0 to 100, resulting in a total score range of 0 to 500.A decrease of 50 points is considered as a minimal clinically important diference . Te IBS Quality of Life (IBS-QoL) comprises 34 IBS-specifc items which divide into 8 variables: health worries, food avoidance, body image, dysphoria, interference with activity, social reactions, sexual activity, and relationships. Te IBS-QoL score will be transformed into a 0-100 scale using the following formula: (the actual raw score - the lowest possible score)/possible score range
  × 100.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT07172139/Prot_000.pdf
  • Informed Consent Form (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT07172139/ICF_001.pdf